CLINICAL TRIAL: NCT04609098
Title: Single Low Dose Tafenoquine to Reduce P. Falciparum Transmission in Mali (NECTAR2)
Acronym: NECTAR2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21905
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Malaria, Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — artenimol; piperaquine; tafenoquine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single blind randomised controlled trial. The treating physician and staff involved with assessing all laboratory outcomes of the study are blinded, but no placebo will be used. The study pharmacist will be unblinded and responsible for randomisation and treatment administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dihydroartemisinin-Piperaquine (DP) (Active Comparator): Subjects will receive Dihydroartemisinin-Piperaquine (DP) once daily for 3 days, and a low dose of 1.66mg/kg, 0.83mg/kg, or 0.415mg/kg. Tafenoquine (TQ) on the first date of DP treatment.
  Interventions: Drug: Dihydroartemisinin/Piperaquine
- DP with 0.415mg/kg Tafenoquine (TQ) (Experimental): Subjects will receive Dihydroartemisinin-Piperaquine (DP) once daily for 3 days, and a single dose of 0.415mg/kg Tafenoquine (TQ) on the first date of DP treatment.
  Interventions: Drug: Dihydroartemisinin/Piperaquine; Drug: Tafenoquine 100mg [Arakoda]
- DP with 0.83 mg/kg TQ (Experimental): Subjects will receive Dihydroartemisinin-Piperaquine (DP) once daily for 3 days, and a single dose of 0.83mg/kg Tafenoquine (TQ) on the first date of DP treatment.
  Interventions: Drug: Dihydroartemisinin/Piperaquine; Drug: Tafenoquine 100mg [Arakoda]
- DP with 1.66mg/kg TQ (Experimental): Subjects will receive Dihydroartemisinin-Piperaquine (DP) once daily for 3 days, and single dose of 1.66mg/kg Tafenoquine (TQ) on the first date of DP treatment.
  Interventions: Drug: Dihydroartemisinin/Piperaquine; Drug: Tafenoquine 100mg [Arakoda]

INTERVENTIONS:
Drug: Dihydroartemisinin/Piperaquine — Tablets containing 40 mg dihydroartemisinin/320 mg piperaquine (Eurartesim, Sigma Tau), administered according to weight as per the manufacturer instructions.
  Other Names: Euartesim
Drug: Tafenoquine 100mg [Arakoda] — Extemporaneous preparation of 1mg/mL Tafenoquine solution, from tablets containing 100mg primaquine (Arakoda, 60degrees pharmaceuticals, DC) dissolved in 100mL water with a non-interacting fruit-flavoured syrup. Solution will be given according to weight as indicated per treatment arm in 5kg bands.
  Other Names: Arakoda
  Arms: DP with 0.415mg/kg Tafenoquine (TQ); DP with 0.83 mg/kg TQ; DP with 1.66mg/kg TQ

SUMMARY:
The purpose of this study is to assess the gametocytocidal and transmission reducing activity of dihydroartemisinin-piperaquine (DP) with and without various low doses of tafenoquine (TQ; 1.66mg/kg, 0.83mg/kg, or 0.415mg/kg). Outcome measures will include infectivity to mosquitoes at 2 and 7 days after treatment, gametocyte density throughout follow-up, and safety measures including haemoglobin density.

DETAILED DESCRIPTION:
Full protocol available on request.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years and ≤ 50 years
* Glucose 6 phosphate dehydrogenase (G6PD) normal status defined by Carestart rapid diagnostic test or the G6PD qualitative test (OSMMR2000)
* Absence of symptomatic falciparum malaria, defined by fever on enrolment
* Presence of P. falciparum gametocytes on thick blood film at a density >16 gametocytes/µL (i.e. ≥ gametocytes recorded in the thick film against 500 white blood cells)
* Absence of other non-P. falciparum species on blood film
* No allergies to study drugs
* No use of antimalarial drugs over the past 7 days (as reported by the participant)
* Hemoglobin ≥ 10 g/dL
* Individuals weighing < = 80 kg
* No evidence of acute severe or chronic disease
* Written, informed consent

Exclusion Criteria:

* Age < 12 years or > 50 years
* Women who are pregnant or lactating
* Blood thick film negative for sexual stages of malaria
* Detection of a non-P. falciparum species by microscopy
* Previous reaction to study drugs / known allergy to study drugs
* Signs of severe malaria, including hyperparasitemia (defined as asexual parasitemia > 100,000 parasites / µL)
* Signs of acute or chronic illness, including hepatitis
* The use of other medication (with the exception of paracetamol and/or aspirin)
* Consent not given
* G6PD-deficiency by Carestart rapid diagnostic test or the OSMMR2000 G6PD qualitative test
* Use of antimalarial drugs over the past 7 days (as reported by the participant)
* The use of other medication (with the exception of paracetamol and/or aspirin)
* Clinically significant illness (intercurrent illness e.g. pneumonia, pre-existing condition e.g. renal disease, malignancy or conditions that may affect absorption of study medication e.g. severe diarrhea or any signs of malnutrition as defined clinically)
* Signs of hepatic injury (such as nausea and/or abdominal pain associated with jaundice) or known severe liver disease (i.e. decompensated cirrhosis, Child Pugh stage B or C)
* Signs, symptoms or known renal impairment
* Clinically significant abnormal laboratory values as determined by history, physical examination or routine blood chemistries and hematology values (laboratory guideline values for exclusion are hemoglobin < 10 g/dL, platelets < 50,000/μl, White Blood Cell count (WBC) < 2000/μl, serum creatinine >2.0mg/dL, or ALT or AST more than 3 times the upper limit of normal for age.
* Family history of diseases leading to QT prolongation or recent treatment with drugs linked to QT prolongation
* Blood transfusion in the last 90 days.
* Consistent with the long half-life of tafenoquine, effective contraception should be continued for 5 half-lives (3 months) after the end of treatment.
* History of psychiatric disorders

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Change in mosquito infectivity assessed through membrane feeding assays (day 7) | 2 days (Days 0 & 7): 7 day span
  The proportion of mosquitoes infected, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 7 post feed, compared to baseline

SECONDARY OUTCOMES:
Change in mosquito infectivity assessed through membrane feeding assays (days 2 and 14) | 3 days (Days 0, 2, & 14): 14 day span
  The proportion of mosquitoes infected, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 2 and 14 post feed, compared to baseline
Mosquito infection density assessed through membrane feeding assays | 4 days (Days 0, 2, 7 & 14): 14 day span
  Mosquito infection density, assessed through membrane feeding and measured as oocyst density in mosquitoes dissected on day 2, 7 and 14 post feed, compared within and between study arms
Mosquito infection prevalence assessed through membrane feeding assays | 4 days (Days 0, 2, 7 & 14): 14 day span
  Mosquito infection prevalence and density, assessed through membrane feeding and measured as oocyst prevalence in mosquitoes dissected on day 2, 7 and 14 post feed, compared within and between study arms
Human infectivity assessed through membrane feeding assays | 4 days (Days 0, 2, 7 & 14): 14 day span
  The proportion of individuals that infect any number of mosquitoes, assessed through membrane feeding and measured as oocyst prevalence/density in mosquitoes dissected on day 2, 7 and 14 post feed, compared within and between study arms
Haemoglobin density | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Haemolysis will be monitored by measuring haemoglobin levels (g/dL) on days 0, 1, 2, 7, 14, 21, and 28 post treatment as part of the clinical assessment.
Methmoglobin density | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Methmoglobin density (g/dL) will be monitored on days 0, 1, 2, 7, 14, 21, and 28 post treatment as part of the clinical assessment.
Aspartate transaminase (AST)/alanine transaminase (ALT) ratio | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Aspartate transaminase (AST)/alanine transaminase (ALT) ratio will be recorded on days 0, 1, 2, 7, 14, 21, and 28 post treatment as part of the clinical assessment.
Blood creatinine level | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Blood creatine level will be recorded on days 0, 1, 2, 7, 14, 21, and 28 post treatment as part of the clinical assessment.
Asexual/sexual stage parasite density | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Asexual/sexual stage parasite density (parasites/microlitre) will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 14, 21, and 28 post treatment.
Asexual/sexual stage parasite prevalence | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Asexual/sexual stage parasite prevalence will be measured by microscopy and by molecular methods on days 0, 1, 2, 7, 14, 21, and 28 post treatment.
Asexual/sexual stage parasite circulation time | 28 days
  Asexual/sexual stage parasite circulation time (days) will be determined from measures of density.
Asexual/sexual stage parasite area under the curve (AUC) | 28 days
  Asexual/sexual stage parasite area under the curve (AUC: Gametocytes per microlitre per day) will be determined from measures of density.
Sexual stage parasite sex ratio | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Gametocyte density will be determined by molecular methods for males and females separately, allowing analysis of sex ratio (proportion of total that is male) on days 0, 1, 2, 7, 14, 21 and 28 post treatment.
Incidence of adverse events | 7 days (Days 0, 1, 2, 7, 14, 21 & 28): 28 day span
  Incidence of adverse events will be monitored at each active (day 0,1,2,7,14,21,28) follow up visit. AE's will also be recorded and acted upon if present at any other time during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Alassane Dicko, PhD, MD, Principal Investigator — Malaria Research and Training Center, Bamako, Mali
Locations (1):
- Malaria Research and Training Centre, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No
Anonymised individual participant data may be shared on a digital repository or upon reasonable request

REFERENCES:
- [Derived] Stone W, Mahamar A, Smit MJ, Sanogo K, Sinaba Y, Niambele SM, Sacko A, Keita S, Dicko OM, Diallo M, Maguiraga SO, Samake S, Attaher O, Lanke K, Ter Heine R, Bradley J, McCall MBB, Issiaka D, Traore SF, Bousema T, Drakeley C, Dicko A. Single low-dose tafenoquine combined with dihydroartemisinin-piperaquine to reduce Plasmodium falciparum transmission in Ouelessebougou, Mali: a phase 2, single-blind, randomised clinical trial. Lancet Microbe. 2022 May;3(5):e336-e347. doi: 10.1016/S2666-5247(21)00356-6. Epub 2022 Mar 23. PMID 35544095